CLINICAL TRIAL: NCT00004005
Title: Irinotecan and 5-Fluorouracil/Leucovorin for Patients With Colorectal Carcinoma and Other Refractory Tumors
Brief Title: Irinotecan Followed By Fluorouracil and Leucovorin in Treating Patients With Stage III or Stage IV Colorectal Carcinoma (Cancer), Other Refractory Carcinoma, or Metastatic Adenoma (Cancer) of Unknown Primary Origin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067216; P30CA021765 (NIH); SJCRH-CACO5; NCI-G99-1554
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2011-10

CONDITIONS: Carcinoma of Unknown Primary; Colorectal Cancer; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific; adenocarcinoma of unknown primary; newly diagnosed carcinoma of unknown primary; recurrent carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, fluorouracil, and leucovorin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with radiation therapy works in treating patients with stage III or stage IV colorectal carcinoma (cancer), other refractory carcinoma (cancer), or metastatic adenocarcinoma (cancer) of unknown primary origin.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with stage IV colorectal carcinoma or other carcinomas treated with irinotecan followed by fluorouracil and leucovorin calcium.
* Determine the disease-free survival of patients with stage III colorectal carcinoma, other refractory carcinomas, or metastatic adenocarcinomas of unknown primary site treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients with stage III colorectal carcinoma (post surgical resection) receive irinotecan IV over 1 hour on days 1-5 and days 8-12. Treatment repeats every 3 weeks for 2 courses. Beginning on week 7, patients receive pelvic irradiation, leucovorin calcium IV over 4 hours, and fluorouracil IV over 5-15 minutes beginning 1 hour into leucovorin calcium infusion on days 1-5. Treatment repeats every 3 weeks for a total of 2 courses. Patients with no evidence of disease may repeat the above 12-week block of chemotherapy without pelvic irradiation up to 4 times over 1 year.

Patients with stage IV colorectal carcinoma, other refractory carcinomas, or metastatic adenocarcinomas of unknown primary site receive the above 12-week block of chemotherapy (irinotecan, fluorouracil, and leucovorin calcium) with pelvic irradiation (if indicated). Pelvic irradiation patients with an unresected primary tumor undergo exploratory surgery 4-5 weeks after completion of radiotherapy, even in the absence of visible tumor regression. Radical resection is attempted to effect local control and control of long term symptoms related to the primary tumor. Patients with complete response (CR) or partial response (PR) after both chemotherapy and surgery repeat the above 12-week block of chemotherapy 3 times over 1 year in the absence of disease progression or unacceptable toxicity. Patients with CR or PR after chemotherapy but no response after surgery receive irinotecan IV over 1 hour on days 1-5 and days 8-12 every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with stable disease (SD) or progressive disease after 2 courses of irinotecan and SD, CR, or PR after surgery receive leucovorin calcium and fluorouracil as above every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically proven previously untreated stage III or stage IV colorectal carcinoma
  * Other carcinomas refractory to standard treatment
  * Metastatic adenocarcinoma of unknown primary site

PATIENT CHARACTERISTICS:

Age:

* Under 25

Performance status:

* ECOG 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Hemoglobin at least 10.0 g/dL
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Albumin greater than 3.0 g/dL
* Bilirubin less than 1.5 mg/dL
* SGOT or SGPT less than 2 times normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 80 mL/min
* Urinalysis normal

Other:

* Blood glucose normal
* Electrolytes normal
* Prior curatively treated childhood cancer allowed
* Weight greater than 10th percentile for height
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 1998-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Response rate
Toxicity
Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Lee Furman, MD, Study Chair — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org